CLINICAL TRIAL: NCT02003976
Title: A Randomized Trial Comparing High Tibial Osteotomy Plus Non-Surgical Treatment and Non-Surgical Treatment Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: The Arthritis Society, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Trevor Birmingham, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-SOG-13-020; MOP-133489 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; high tibial osteotomy; gait analysis; muscular strength; body composition; magnetic resonance imaging; biological markers
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Surgical Treatment plus HTO (Experimental): The optimized non-surgical treatment program consists of medications, physiotherapy and nutritional seminars. The 12-week program will include an assessment by a primary care physician, physiotherapist and orthopaedic surgeon, one supervised physiotherapy session per week, one body recomposition session per week, and a home program. After the 12-week program is completed, patients randomized to this group will undergo a medial opening wedge high tibial osteotomy (HTO). They will continue with their home program and will be followed up for 2 years after baseline.
  Interventions: Procedure: Medial Opening Wedge High Tibial Osteotomy (HTO); Other: Non-Surgical Treatment Program
- Non-Surgical Treatment (Active Comparator): The optimized non-surgical treatment program consists of medications, physiotherapy and nutritional seminars. The 12-week program will include an assessment by a primary care physician, physiotherapist and orthopaedic surgeon, one supervised physiotherapy session per week, one body recomposition session per week, and a home program. After the 12-week program is completed, patients randomized to this group will continue with their home program and will be followed up for 2 years after baseline.
  Interventions: Other: Non-Surgical Treatment Program

INTERVENTIONS:
Procedure: Medial Opening Wedge High Tibial Osteotomy (HTO) — A lower limb realignment surgery to redistribute load away from the most affected portion of the knee.
  Arms: Non-Surgical Treatment plus HTO
Other: Non-Surgical Treatment Program — A 12-week optimized non-surgical treatment program consisting of medication, physiotherapy and nutritional seminars.

SUMMARY:
The purpose of this study is to compare patients with knee osteoarthritis (OA) receiving optimized non-surgical treatment plus surgical realignment of the tibia, or optimized non-surgical treatment only. We hypothesize that outcomes assessed at 12 and 24 months follow-up will suggest favourable changes in patients undergoing surgical realignment when compared to patients receiving non-surgical treatment only.

DETAILED DESCRIPTION:
This two groups, parallel design randomized controlled trial will compare patients with medial compartment knee OA and varus alignment receiving optimized non-surgical treatment plus High Tibial Osteotomy (HTO) to similar patients receiving optimized non-surgical treatment only. All participants will receive non-surgical treatment that will be individualized to the patient and include medications, physiotherapy and nutritional seminars. The non-surgical treatment will include supervised physiotherapy and nutritional seminars once per week for 12 weeks, will be accompanied and followed by a home program, and follow-up appointments for potential modification every three months for the duration of the study. Participants randomized to surgery will also undergo medial opening wedge HTO after 12 weeks of optimized non-surgical treatment. Both groups will follow the same schedule of clinic visits throughout the 24 month follow-up period. MRI-derived measures of articular cartilage morphology, biological markers of articular cartilage degradation and synthesis, gait biomechanics and patient-reported outcomes will be assessed at baseline, 12 and 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject either:

   1. 25-55 years old?
   2. Older than 55 but still active (ex. physical labour, regular recreational activities)?
2. Does this subject present with varus alignment? (Based on hip to ankle x-rays).
3. Does this subject have clinical Knee OA? (MAA <-2° on full limb standing AP) according to the Altman classification primarily involving the medial compartment of the knee?
4. Patient is a good candidate for high tibial osteotomy and will be receiving a PEEK plate, or if receiving an alternate plate, agrees to have the plate removed prior to 1 year postoperative.

Exclusion Criteria:

1. Has this subject had a previous HTO or joint replacement in either limb?
2. Is this subject likely to undergo bilateral HTO within the 2 year follow up period?
3. Does this subject have an unstable knee or ligament?
4. Does this subject have inflammatory or infectious arthritis of the knee?
5. Radiographic disease too advanced for HTO (ie. diffuse lateral compartment, patellofemoral joint OA and/or severe enough disease to suggest that joint replacement is the better surgical option) and/or Kellgren and Lawrence grade 4.
6. The subject's disease is not advanced enough (symptomatically or radiographically) to warrant HTO.
7. Does this subject have a major medical illness with life expectancy <2 years or with an unacceptably high operative risk?
8. Does this subject have a major neurological deficit that would affect gait?
9. Is this subject possibly pregnant or planning pregnancy?
10. Is this subject unable to read English?
11. Does this subject have a psychiatric illness that limits informed consent?
12. Is the subject unlikely to comply with study protocol?

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
MRI articular cartilage morphology | Change from baseline to 24 months post operative
  3 Tesla MRI measure of medial tibiofemoral articular cartilage thickness

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from baseline to 24 months post operative
  Patient-reported outcome measure. 5 subdomains: pain, symptoms, activities of daily living, sport and recreation, quality of life
Western Ontario Meniscal Evaluation Tool (WOMET) | Change from baseline to 24 months post operative
  Patient-reported outcome measure. Assesses health-related quality of life (HRQoL) in patients with meniscal tears. 3 dimensions: physical symptoms, sports/recreation/work/lifestyle, emotions
Biological Markers of Disease Progression | Baseline, 12 and 24 months post operative
  Synovial fluid, serum and urine biological markers
Numeric Rating Scale for Pain | Baseline, 12 and 24 months post operative
  Patient-reported outcome measure. Assesses patient's pain. 0 (no pain) - 10 (worst possible pain)
Gait Biomechanics | Baseline, 12 and 24 months post operative
  Knee frontal, sagittal and transverse plane kinematics and kinetics tested during level walking in a motion analysis laboratory. The measure of most interest is the peak external knee adduction moment during stance phase of walking.
Isometric Strength Testing | Baseline, 12 and 24 months post operative
  Isometric quadriceps and hamstrings strength tested using an isokinetic dynamometer.
Intermittent and Constant Osteoarthritis Pain Index (ICOAP) | Change from baseline to 24 months post operative
  Patient-reported outcome measure. Assesses pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain. 3 domains: intermittent pain, constant pain, total pain
Short-Form 12 (SF12) | Change from baseline to 24 months post operative
  Patient-reported outcome measure. Self-reported outcome measure assessing the impact of health on an individual's everyday life
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Change from baseline to 24 months post operative
  Patient-reported outcome measure. 3 sub domains: pain, symptoms, function

OTHER OUTCOMES:
Cost-effectiveness questionnaires | Baseline and every 3 months from baseline up to 24 months post operative
  Collection of accumulated direct and indirect costs related to the intervention incurred over the study period as reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor B Birmingham, PT, PhD, Principal Investigator — Western University; J R Giffin, MD, Principal Investigator — Western University
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birmingham TB, Primeau CA, Moyer RF, Bryant DM, Ma J, Leitch KM, Wirth W, Degen R, Getgood AM, Litchfield RB, Willits KR, Eckstein F, Giffin JR. High Tibial Osteotomy for Medial Compartment Knee Osteoarthritis : A Randomized Trial With Parallel Preference Arm. Ann Intern Med. 2025 Sep;178(9):1238-1248. doi: 10.7326/ANNALS-25-00920. Epub 2025 Jul 29. PMID 40720836